CLINICAL TRIAL: NCT01957865
Title: Development of a Real-Time Antiretroviral Therapy Adherence Intervention in Uganda
Brief Title: Real-Time Antiretroviral Therapy Adherence Intervention in Uganda
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Mbarara University of Science and Technology (Other)
Responsible Party: Principal Investigator, Jessica Haberer, MD, Assistant Professor of Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: R34MH100940-01 (NIH)
Record Dates: First submitted 2013-09-25; First posted 2013-10-08 (Estimated); Results first posted 2016-11-10 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2016-11

CONDITIONS: HIV/AIDS; Adherence
Keywords: HIV/AIDS; adherence; real time monitoring; SMS; mHealth; social support
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Fixed SMS, real-time monitoring (Experimental): SMS will be sent daily for one month, then weekly for two months. Participants will have real-time adherence monitoring and social supporters will be notified of gaps in adherence of 48+ hours in the last six months of the study.
  Interventions: Device: Fixed SMS, real-time monitoring
- Triggered SMS, real-time monitoring (Experimental): Participants will have real-time adherence monitoring and social supporters will be notified of gaps in adherence of 48+ hours in the last six months of the study.
  Interventions: Device: Triggered SMS, real-time monitoring
- control (No Intervention): Real-time adherence monitoring only (no SMS)

INTERVENTIONS:
Device: Fixed SMS, real-time monitoring — SMS reminders will be sent daily for one month, then weekly for two months, then as needed for missed doses to encourage adherence. The Wisepill system will automatically capture and report each time the device is opened as a proxy for the participant's adherence.
  Other Names: Wisepill
  Arms: Fixed SMS, real-time monitoring
Device: Triggered SMS, real-time monitoring — SMS reminders will be sent as needed for missed doses to encourage adherence. The Wisepill system will automatically capture and report each time the device is opened as a proxy for the participant's adherence.
  Other Names: Wisepill
  Arms: Triggered SMS, real-time monitoring

SUMMARY:
Development of Real-Time Antiretroviral Therapy Adherence Intervention in Uganda (The Wisepill Study).

DETAILED DESCRIPTION:
In this study, the investigators propose to develop a real-time adherence intervention based on SMS (i.e., text messages), wireless adherence monitoring (with the Wisepill device), and engagement of social support that is tailored to rural sub-Saharan Africa. The investigators will build on research by others who have shown SMS reminders improve adherence and viral suppression in Kenya, albeit with relatively small effect sizes and suboptimal virologic failure rates even in the intervention arm. Moreover, little is known about which patients benefit from SMS, why they benefit, and what can be done to further improve adherence and treatment success rates. Understanding the mechanisms of effect will make it possible to design and test evidence-based interventions with the highest likelihood for efficacy.

In a cohort of HIV-infected individuals starting ART and being monitored with Wisepill, the investigators will test 1) daily SMS reminders, 2) weekly SMS reminders, 3) SMS reminders linked to real-time detection of missed doses, and 4) SMS reminders plus SMS notifications of 48+hour gaps in adherence to members of social support networks. The investigators will conduct qualitative interviews to learn the experiences of participants and members of their social support networks with the different types of SMS. This staged approach will allow us to fully understand and compare the additive effects and acceptability of SMS-based interventions. The investigators will also determine behavioral effect mechanisms, as well as compare the impact of each type of SMS with a control population receiving only Wisepill monitoring on adherence and HIV RNA.

ELIGIBILITY:
Wisepill Participants:

Inclusion Criteria:

* HIV-infected
* Initiating ART within the next two weeks
* Age 18 years and older
* Owns a cell phone for personal use and has reliable cellular phone reception at home on a network supported by the technology used in this study
* Lives in the Mbarara District (i.e, within 20 km of the ISS Clinic)
* Has at least one person who could be named as a social supporter(see criteria below).

Exclusion Criteria:

* Unable to use SMS
* Unwilling to receive SMS reminders
* Severe mental condition limiting the ability to provide consent
* Cellular phone reception is not reliable

Social supporters (i.e., recipients of the SMS notifications for Wisepill participants in the intervention arms):

Inclusion criteria:

* Knows Wisepill participant has HIV
* Age 18 years or older
* Reports having provided social support to the intervention participant at least once
* Own a cell phone for personal use and have reliable cellular phone reception at home on a network supported by the technology used in this study
* Lives in the Mbarara District

Exclusion criteria:

* Unable to use SMS
* Unwilling to receive SMS notifications regarding interruptions in the intervention participant's adherence
* Severe mental condition limiting the ability to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2013-09; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Haberer, MD, MS, Principal Investigator — Massachusetts General Hospital; Angella Musiimenta, PhD, Principal Investigator — Mbarara University of Science and Technology
Locations (1):
- Mbarara Immune Suppression Syndrome(ISS) Clinic, Mbarara, Mbarara District, Uganda

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be available at the end of the study upon request.

REFERENCES:
- [Derived] Musiimenta A, Atukunda EC, Tumuhimbise W, Haberer JE. Resilience after withdrawing a technology-based medication adherence support intervention from people living with HIV in rural Uganda. AIDS Care. 2018 Aug;30(sup5):S89-S96. doi: 10.1080/09540121.2018.1510107. Epub 2019 Jan 9. PMID 30626191
- [Derived] Musiimenta A, Atukunda EC, Tumuhimbise W, Pisarski EE, Tam M, Wyatt MA, Ware NC, Haberer JE. Acceptability and Feasibility of Real-Time Antiretroviral Therapy Adherence Interventions in Rural Uganda: Mixed-Method Pilot Randomized Controlled Trial. JMIR Mhealth Uhealth. 2018 May 17;6(5):e122. doi: 10.2196/mhealth.9031. PMID 29773527
- [Derived] Haberer JE, Musiimenta A, Atukunda EC, Musinguzi N, Wyatt MA, Ware NC, Bangsberg DR. Short message service (SMS) reminders and real-time adherence monitoring improve antiretroviral therapy adherence in rural Uganda. AIDS. 2016 May 15;30(8):1295-300. doi: 10.1097/QAD.0000000000001021. PMID 26760452

RESULTS

PARTICIPANT FLOW:
Groups:
- Fixed SMS, Real-time Monitoring: SMS were sent daily for one month, then weekly for two months and then after missed doses for the remainder of the study. Participants had real-time adherence monitoring and social supporters were notified of gaps in adherence of 48+ hours in the last six months of the study.
- Triggered SMS, Real-time Monitoring: SMS were sent for missed doses throughout the study. Participants had real-time adherence monitoring and social supporters were notified of gaps in adherence of 48+ hours in the last six months of the study.
Period: Overall Study
Arm/Group | Fixed SMS, Real-time Monitoring | Triggered SMS, Real-time Monitoring | Control
Started | 21 | 20 | 22
Completed | 21 | 18 | 19
Not Completed | 0 | 2 | 3
Not completed — Found HIV negative | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fixed SMS, Real-time Monitoring | Triggered SMS, Real-time Monitoring | Control | Total
Number analyzed (Participants) | 21 | 20 | 22 | 63
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 33 [28 to 40] | 33 [26 to 35] | 27 [24 to 32] | 30 [25 to 35]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 7 | 19 | 41
  Male | 6 | 13 | 3 | 22
Region of Enrollment [Number; unit: participants]
  Uganda | 21 | 20 | 22 | 63
Median CD4 count [Median (Inter-Quartile Range); unit: cells/mm^3] | 309 [241 to 385] | 291 [213 to 350] | 382 [249 to 457] | 309 [231 to 397]

OUTCOME MEASURES:

1. Primary Outcome: Antiretroviral Therapy (ART) Adherence Levels
Description: ART adherence in each study arms. Adherence is measured by the Wisepill real-time adherence monitor and calculated as the number of monitor opening signals received divided by the number of monitor opening signals expected, capped at 100%.
Time Frame: real time (for 9 months)
Population: The participant found to be HIV negative was not included in the analysis.
Measure: Mean (Standard Deviation); unit: Percent adherence
Groups:
- Fixed SMS, Real-time Monitoring: Fixed SMS, real-time monitoring: SMS reminders were sent daily for one month, then weekly for two months, then as needed for missed doses to encourage adherence. Participants had real-time adherence monitoring and social supporters were notified of gaps in adherence of 48+ hours in the last six months of the study.
  The Wisepill system automatically captured and reported each time the device was opened as a proxy for the participant's adherence.
- Triggered SMS, Real-time Monitoring: Triggered SMS, real-time monitoring: SMS reminders were sent as needed for missed doses to encourage adherence. Participants had real-time adherence monitoring and social supporters were notified of gaps in adherence of 48+ hours in the last six months of the study.
  The Wisepill system automatically captured and reported each time the device was opened as a proxy for the participant's adherence.
Arm/Group | Fixed SMS, Real-time Monitoring | Triggered SMS, Real-time Monitoring | Control
Number analyzed (Participants) | 21 | 20 | 21
Percent adherence | 91 (9) | 79 (18) | 79 (22)
Statistical Analysis 1: Comparison: Fixed SMS, Real-time Monitoring vs Triggered SMS, Real-time Monitoring vs Control; In an intention-to-treat analysis, percentage doses taken each month were compared by linear generalized estimating equations (GEEs); more than 48-h and more than 96-h lapses in dosingwere compared by Poisson GEE regression; Test type: Superiority or Other; p < 0.05, Linear and Poisson regressions

2. Secondary Outcome: HIV RNA Suppression
Description: HIV RNA suppression (<100 copies/ml) in each study arm
Time Frame: After month 9
Population: Note: Missing data equals lack of suppression. The participant found to be HIV negative was not included in the analysis.
Measure: Number; unit: number of participants
Arm/Group | Fixed SMS, Real-time Monitoring | Triggered SMS, Real-time Monitoring | Control
Number analyzed (Participants) | 21 | 20 | 21
number of participants | 20 | 15 | 19
Statistical Analysis 1: Comparison: Fixed SMS, Real-time Monitoring vs Triggered SMS, Real-time Monitoring vs Control; HIV RNA suppression (<100 copies/ml) was compared among study arms by Fisher's exact test; Test type: Superiority or Other; p < 0.05, Fisher's exact test

ADVERSE EVENTS:
Time Frame: 1 year, 9 months
Groups:
- Fixed SMS, Real-time Monitoring: SMS were sent daily for one month, then weekly for two months. Participants had real-time adherence monitoring and social supporters were notified of gaps in adherence of 48+ hours in the last six months of the study.
  Fixed SMS, real-time monitoring: SMS reminders were sent daily for one month, then weekly for two months, then as needed for missed doses to encourage adherence. The Wisepill system automatically captured and reported each time the device is opened as a proxy for the participant's adherence.
- Triggered SMS, Real-time Monitoring: Participants had real-time adherence monitoring and social supporters were notified of gaps in adherence of 48+ hours in the last six months of the study.
  Triggered SMS, real-time monitoring: SMS reminders were sent as needed for missed doses to encourage adherence. The Wisepill system automatically captured and reported each time the device is opened as a proxy for the participant's adherence.
Arm/Group | Fixed SMS, Real-time Monitoring | Triggered SMS, Real-time Monitoring | Control
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/20 | 0/22
Other Adverse Events (participants affected / at risk) | 0/21 | 0/20 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No